CLINICAL TRIAL: NCT06714903
Title: Multi-omics Study of Intestinal Microecology in Patients with Colorectal Cancer Related to Immunotherapy
Brief Title: Effect of Gut Microbiota and Its Metabolites on the Efficacy of Immunotherapy in Metastatic Colorectal Cancer
Status: Recruiting | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-HS-147
Record Dates: First submitted 2024-12-02; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Neoplasms Malignant
Keywords: Metastatic colorectal cancer; Immunotherapy; Gut microbiota; Prognosis; Metabolism
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — blood samples and stool samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Experimental group: sintilimab + fruquintinib
  Interventions: Other: treatment option-sintilimab plus fruquintinib
- Control group: fruquintinib
  Interventions: Other: treatment option-fruquintinib alone

INTERVENTIONS:
Other: treatment option-sintilimab plus fruquintinib — sintilimab plus fruquintinib
  Groups: Experimental group
Other: treatment option-fruquintinib alone — fruquintinib alone
  Groups: Control group

SUMMARY:
The purpose of this observational study is to understand the effect of gut microbiota on the efficacy of immunotherapy in patients with metastatic colorectal cancer and to explore the specific mechanisms of this process. In this way, it provides new ideas for the clinical treatment of colorectal cancer.

DETAILED DESCRIPTION:
This study is a single-center, prospective, observational study. This study plans to enroll 50 patients with mCRC who received immunotherapy. Stool and blood samples were collected from patients with mCRC before receiving immunotherapy (baseline) and after one cycle of immunotherapy and stored immediately in a -80°C freezer. Six months after treatment with a PD-1 inhibitor in combination with fruquintinib, patients with mCRC were evaluated radiographically according to the modified RECIST1.1 criteria for immunotherapy (iRECIST) and were divided into responsive and non-responsive groups.

In this study, we intend to use metagenomic sequencing to screen the key intestinal microbiota that affect the efficacy of PD-1 inhibitors and predict their possible functional pathways in patients with metastatic colorectal cancer receiving anti-PD-1 immunotherapy. Then, proteomics and metabolomics methods were used to screen differential proteins and metabolites, and the correlation analysis with key intestinal microbiota was carried out, and the efficacy of immunotherapy in patients with mCRC was evaluated. Finally, the above findings were verified in animal models, and then the specific mechanism of intestinal microbiota affecting the efficacy of PD-1 inhibitors was explained by taking the changes in body metabolism and immunity as the starting point.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and pathological diagnosis of metastatic colorectal cancer
* 35-75 years old (both ends inclusive)
* complete clinical information
* signed informed consent

Exclusion Criteria:

* combined with severe respiratory and circulatory diseases
* combined with other malignant tumors
* recent severe active bleeding, uncontrolled active infection or active peptic ulcer
* moderate to severe renal insufficiency
* other circumstances that are judged by the investigator to be unsuitable for participating in this study

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 50 patients with metastatic colorectal cancer who received immunotherapy from the First Hospital of Jilin University from 2024 to 2026 were included
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of efficacy | six months after treatment
  Six months after treatment with a PD-1 inhibitor in combination with fruquintinib, patients with mCRC were evaluated radiographically according to the modified RECIST1.1 criteria for immunotherapy (iRECIST) and were divided into responsive and non-responsive groups. Patients are classified as responders if they achieve an objective response (complete or partial response or stable disease for at least 6 months), while patients are classified as non-responders if they have progressed on treatment or have stable disease for less than 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Nan Zhang, Study Director — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided